CLINICAL TRIAL: NCT00077688
Title: A Phase 2 Multicenter Evaluation of the Safety and Efficacy of TOCOSOL(TM) Paclitaxel (S-8184 Paclitaxel Injectable Emulsion) in Patients With Metastatic or Locally Advanced, Unresectable Transitional Cell Carcinoma of the Urothelium
Brief Title: TOCOSOL(TM) Paclitaxel in Metastatic or Locally Advanced Unresectable Transitional Cell Carcinoma of the Urothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SON-8184-1073
Record Dates: First submitted 2004-02-10; First posted 2004-02-16 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms; Carcinoma, Transitional Cell
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms; Carcinoma, Transitional Cell

INTERVENTIONS:
Drug: TOCOSOL Paclitaxel

SUMMARY:
Phase 2B, multicenter study evaluating the safety and efficacy of weekly TOCOSOL Paclitaxel in taxane-naive patients receiving second line chemotherapy for metastatic or locally advanced, unresectable transitional cell carcinoma of the urothelium

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of transitional cell carcinoma (TCC) of the urothelium including bladder, renal pelvis, ureter, or urethra
* Stage IV disease
* One and only one prior systemic cytotoxic chemotherapy regimen administered as adjuvant or neoadjuvant chemotherapy or to treat locally advanced or metastatic disease
* Adequate hematologic function (ANC >/= 1500 cells/mm3 & platelet count >/= 100,000/mm3)
* Serum creatinine </= 2.0 mg/dL
* Total bilirubin </= 1.5 mg/dL
* SGOT & SGPT </= 3 times upper limit of institutional normal values
* PT (INR) & PTT within institutional lab normal range
* Karnofsky performance status of 60-100%
* At least one unidimensionally measurable lesion, suitable for radiographic evaluation of disease response, consistent with RECIST criteria
* Signed IRB/EC approved Informed Consent
* Life expectancy of at least 12 weeks
* 18 years of age or older
* Fully recovered from any previous surgery
* Not pregnant and willing to use a medically effective form of contraception during periods of chemotherapy treatment (both males and and females)
* Agree not to take vitamin E supplementation while receiving study medication
* Willing to participate in requested follow-up evaluations
* Willing to permit treating physicians to provide information to Sonus regarding disease status and survival for 2 years after first dose of study drug

Exclusion Criteria:

* Prior taxane-containing chemotherapy including Taxol(R) (paclitaxel) or generic equivalent, or Taxotere(R) (docetaxel)
* Peripheral neuropathy NCI-CTC grade 2 or greater
* Wide-field radiation, cytotoxic chemotherapy or hormonal therapy within 4 weeks of first dose, or mitomycin or nitrosoureas within 6 weeks of first dose, of study drug
* An investigational agent within 4 weeks of first dose of study drug
* Concurrent anticonvulsants known to induce P450 isoenzymes
* Patients who are pregnant or lactating
* A history of carcinoma of another primary site (other than non-melanoma skin cancers or carcinoma-in-situ of the cervix) within the previous 5 years, unless metastatic disease has been biopsied and documented to be TCC
* Bone metastasis, effusions, ascites or elevated tumor markers as the only evidence of metastatic TCC
* Brain metastasis
* Active bowel obstruction
* Active, serious infection or other serious medical problems (other than TCC) likely to impair completion of the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44
Dates: Start 2003-11; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Objective response rate

SECONDARY OUTCOMES:
Time to treatment failure
Time to progression
Progression free survival
Overall survival at 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Maryland Medical Center/Greenbaum Cancer Center, Baltimore, Maryland
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington